CLINICAL TRIAL: NCT04640987
Title: Phase 1/1b Study of T-allo10 Infusion After HLA-Partially Matched Related or Unrelated TCR αβ+ T-cell/ CD19+ B-cell Depleted Allogeneic Hematopoietic Stem Cell Transplantation (αβ Depleted-HSCT) in Children and Young Adults Affected by Hematologic Malignancies
Brief Title: Stem Cell Transplant From Donors After Alpha Beta Cell Depletion in Children and Adults With T-allo10 Cells Addback
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Porteus, Matthew, MD (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Principal Investigator, Alice Bertaina, Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-58549; BMT 367 - T-allo10 Alpha Beta (Other: Stanford University)
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): The participant will undergo a alpha-beta depleted stem cell transplant using donor cells. The participant's cells will then be manipulated via a T-allo10 cell addback to reach a dose level of 1 X 10^5/kg
  Interventions: Biological: Allogeneic Stem Cell Transplant; Device: CliniMACS Prodigy System; Drug: T-allo10 cells addback
- Cohort 2 (Experimental): The participant will undergo a alpha-beta depleted stem cell transplant using donor cells. The participant's cells will then be manipulated via a T-allo10 cell addback to reach a dose level of 3 X 10^5/kg
  Interventions: Biological: Allogeneic Stem Cell Transplant; Device: CliniMACS Prodigy System; Drug: T-allo10 cells addback
- Cohort 3 (Experimental): The participant will undergo a alpha-beta depleted stem cell transplant using donor cells. The participant's cells will then be manipulated via a T-allo10 cell addback to reach a dose level of 1 X 10^6/kg
  Interventions: Biological: Allogeneic Stem Cell Transplant; Device: CliniMACS Prodigy System; Drug: T-allo10 cells addback

INTERVENTIONS:
Biological: Allogeneic Stem Cell Transplant — The allogeneic stem cell transplant involves transferring the stem cells from a healthy person (donor) to the participant via infusion.
Device: CliniMACS Prodigy System — Device used for production of T-allo10 cells.
Drug: T-allo10 cells addback — T-allo10 cells are made by manipulating the participant's stem cell donor's white blood cells (CD4+ T cells) in the presence of their (participant's) CD14+ monocytes.

SUMMARY:
The purpose of this study is to determine the safety of a cell therapy, T-allo10, after αβdepleted-HSCT in the hopes that it will boost the adaptive immune reconstitution of the patient while sparing the risk of developing severe Graft-versus-Host Disease (GvHD).

The primary objective of Phase 1a is to determine the recommended Phase 2 dose (RP2D) administered after infusion of αβdepleted-HSCT in children and young adults with hematologic malignancies.

A Phase 1b extension will occur after dose escalation, enrolling at the RP2D for the T-allo10 cells determined in the Phase 1 portion to evaluate the safety and efficacy of infusion of T-allo10 after receipt of αβdepleted-HSCT. Additionally, Phase 1b aims to explore improvements in immune reconstitution.

All participants on this study must be enrolled on another study: NCT04249830

ELIGIBILITY:
Inclusion Criteria prior to enrollment:

* 1. Age > 1 months (with minimum weight of 10 Kg) and < 45 years.
* 2. Patients deemed eligible for allogeneic HSCT under the originating study, NCT 04249830
* 3. Patients with life-threatening hematological malignancies for which HSCT has been recommended:

  1. High-risk ALL in 1st CR, ALL in 2nd or subsequent CR;
  2. High-risk AML in 1st CR, AML in 2nd or subsequent CR;
  3. Myelodysplastic syndrome;
  4. JMML (Juvenile myelomonocytic leukemia);
  5. Non-Hodgkin lymphomas in 2nd or subsequent CR;
  6. Other hematologic malignancies eligible for stem cell transplantation per institutional standard.
* 4. All subjects ≥ 18 years of age must be able to give informed consent, or adults lacking capacity to consent must have a LAR available to provide consent. For subjects <18 years old their LAR (i.e. parent or guardian) must give informed consent. Pediatric subjects will be included in age appropriate discussion and verbal assent will be obtained for those > 7 years of age, when appropriate.

Inclusion criteria prior to T-allo10 infusion:

1. Patient already received αβdepleted-HSCT and has myeloid engraftment.
2. Absence of active grade II aGvHD requiring >0.5 mg/Kg of steroids or any diagnosis of grade III/IVaGvHD.

Exclusion Criteria prior to MNC collection for Tallo-10 manufacturing.:

1. Not eligible to receive HSCT on NCT04249830
2. Received another investigational agent within 30 days of enrollment.
3. Pregnancy (positive serum or urine beta-HCG) within 7 days of MNC donation.
4. Patient or donor is not willing or able to undergo an additional non-mobilized apheresis for collection of MNC prior to donation of cells for participation in NCT04249830.

Ages: 1 Month to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of T-allo10 in Phase 1a | Up to 28 days after infusion of T-allo10 for each dosing cohort and Day +60 (+/- 10 days) after αβdepleted-HSCT
  RP2D was determined by testing 3 different escalating doses (1x10^5, 3x10^5 and 1x10^6 cells/Kg recipient body weight) in dose escalation cohorts 1 to 3 with 3 to 6 participants each. RP2D reflects the acceptable dose levels that did not cause a Dose-Limiting Toxicity (DLT) in ≥33% of participants and resulted in success with response in >83% of participants. DLTs were defined as Grade IV aGvHD post T-allo10 infusion; any grade 3 or 4 related TEAE; any grade 3 or 4 suspected AE. Success with response was defined as achieving CD4+ IR by Day +60 (+/- 10 days) after αβdepleted-HSCT.
Number of participants with absence of dose-limiting toxicity (DLT) | Assessed at 28 days (after infusion of T-allo10)
  Grade IV aGvHD post T-allo10 infusion; any grade 3 or 4 related treatment emergent adverse events (TEAE); any grade 3 or 4 suspected AE
Number of participants who reach immune reconstitution (IR) threshold | Up to Day 60 (+/- 10 days) after αβdepleted-HSCT
  IR (a surrogate of reduced risk of leukemia recurrence) is defined reaching the threshold of 50CD3+CD4+T-cells/µl by Day+60 (+/-10days).

SECONDARY OUTCOMES:
Number of participants with ≥grade 3 adverse event related to T-allo10 infusion | Through 1 year after αβdepleted-HSCT
Number of participants with grade II-IV aGvHD | Assessed at day 90 and day 180 after αβdepleted-HSCT
  Cumulative incidence of acute GvHD (graded as II-IV using the Magic criteria)
Number of participants with grade III-IV aGvHD | Assessed at day 90 and day 180 after αβdepleted-HSCT
  Cumulative incidence of acute GvHD (graded as III-IV using the Magic criteria)
Number of participants with cGvHD | Assessed at 1 year after αβdepleted-HSCT
  Chronic GvHD is graded according to the NIH Consensus Conference criteria
Number of participants who achieved leukemia-free survival | Assessed at 1 year after αβdepleted-HSCT
  Leukemia-free survival defined as at the time of enrollment to disease relapse or death from any cause.
Number of participants with disease relapse | Assessed at 1 year after αβdepleted-HSCT
  Disease relapse is defined as the return of signs and symptoms of a disease after a remission.
Non-relapse mortality | Assessed at Day 90, 1 year after αβdepleted-HSCT
  Non-relapse mortality is defined as death not preceded by recurrent primary malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bertaina, MD, PhD, Principal Investigator — Professor of Pediatrics, Stem Cell Transplantation
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No